CLINICAL TRIAL: NCT02953561
Title: An Open-Label Phase Ib/II Study of Avelumab in Combination With 5-Azacytidine (Vidaza) for the Treatment of Patients With Refractory/Relapsed Acute Myeloid Leukemia
Brief Title: Avelumab and Azacitidine in Treating Patients With Refractory or Relapsed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PDOL request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0444; NCI-2016-01924 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0444 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — avelumab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (azacitidine, avelumab) (Experimental): Patients receive azacitidine SC or IV over 10-40 minutes on days 1-7 or on days 1-5 and 8-9. Patients also receive avelumab IV over 60 minutes on days 1 and 14 for 4 courses (or until complete response) and on day 1 for subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Drug: Azacitidine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase Ib/II trial studies the best dose and side effects of avelumab when given together with azacitidine and to see how well they work in treating patients with acute myeloid leukemia that is not responding to treatment or has come back. Monoclonal antibodies, such as avelumab, may interfere with the ability of cancer cells to grow and spread. Azacitidine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving avelumab and azacitidine may work better in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of avelumab in combination with azacitidine (5-azacytidine) in patients with refractory/relapsed acute myeloid leukemia (AML). (Phase IB)

II. To determine the overall response rate (ORR) defined as complete remission (CR)/complete remission with incomplete platelet recovery (CRp)/complete remission with incomplete count recovery (CRi)/partial remission (PR)/hematologic improvement (HI)/morphologic leukemia free state (MLFS) of avelumab in combination with 5-azacytidine in patients with refractory/relapsed AML. (Phase II

SECONDARY OBJECTIVES:

I. To determine the number of patients achieve > 50% reduction in blasts on therapy with this combination.

II. To determine the duration of response, disease-free survival (DFS), and overall survival (OS) of patients with refractory/relapsed AML treated with this combination

TERTIARY OBJECTIVES:

I. To study immunological and molecular features at baseline and at predefined time-points on-therapy with avelumab and azacytidine in the peripheral blood and bone marrow to include quantify immune ligand expression by the AML blasts and AML stromal components (myeloid-derived suppressor cells [MDSCs] and mesenchymal stem cells [MSCs]) including 4-1BBL, ICOSL, PD-L1, PD-L2, OX-40L, CD137L.

II. To study immunological and molecular features at baseline and at predefined time-points on-therapy with avelumab and azacytidine in the peripheral blood and bone marrow to determine the quantitative expression of positive and negative co-stimulatory molecules on individual T-lymphocyte subsets including 4-1BB, CTLA-4, ICOS, PD-1, OX40, LAG-3 and TIM-3.

III. To study immunological and molecular features at baseline and at predefined time-points on-therapy with avelumab and azacytidine in the peripheral blood and bone marrow to identify the immunophenotype of tumor-infiltrating T-lymphocytes (TILs) pre- and post-therapy with the combination: CD8+, CD4+ effector, or CD4+ regulatory.

IV. To develop a micro-array based gene expression profile (GEP) predictor of response to anti-PDL1 and epigenetic therapy in AML.

V. To determine the correlation of responses to the combination with baseline cytogenetic and molecular abnormalities

OUTLINE: This is a phase Ib, dose-escalation study of avelumab followed by a phase II study

Patients receive azacitidine subcutaneously (SC) or intravenously (IV) over 10-40 minutes on days 1-7 or on days 1-5 and 8-9. Patients also receive avelumab IV over 60 minutes on days 1 and 14 for 4 courses (or until complete response) and on day 1 for subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity

After completion of study treatment, patients are followed up every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML who are refractory (up to salvage 2) or relapsed (up to 2nd relapse); for patients with prior myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) or myeloproliferative neoplasm (MPN) who transformed to AML, therapy received for MDS, CMML, or MPN is NOT considered as prior therapy for AML
* Prior therapy with hydroxyurea, chemotherapy, biological or targeted therapy (e.g. FLT3 inhibitors, other kinase inhibitors), or hematopoietic growth factors is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 1.5 times upper limit of normal (x ULN) (=< 3 x ULN if considered to be due to leukemic involvement or Gilbert's syndrome)
* Aspartate aminotransferase or alanine aminotransferase =< 2.5 x ULN (=< 5.0 x ULN if considered to be due to leukemic involvement)
* Estimated creatinine clearance >= 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
* Patients must provide written informed consent
* In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of 5-azacytidine and avelumab will be at least 14 days OR at least 5 half-lives for cytotoxic/noncytotoxic agents, whichever is longer; the toxicity from prior therapy should have resolved to grade =< 1, however alopecia and sensory neuropathy grade =< 2 is acceptable; the half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochures, or drug-administration manuals) and will be documented in the protocol eligibility document; use of hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and will not require a washout; concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted; patients with CNS disease or leukemic brain metastasis must have been treated locally and be clinically stable for at least 2 weeks prior to enrollment and have no ongoing neurological symptoms that are related to the CNS disease (sequelae that are a consequence of the treatment of the CNS disease are acceptable)
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment; males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment; adequate methods of contraception include:

  * Total abstinence when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening); for female patients on the study, the vasectomized male partner should be the sole partner for that patient
  * Combination of any of the two following (a+b or a+c or b+c)

    * a. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
    * b. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * c. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository In case of use of oral contraception, women should have been stable on the same pill before taking study treatment
  * Note: oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential

Exclusion Criteria:

* Patients with a known allergy or hypersensitivity to avelumab, 5-azacytidine, or any of their components; known severe hypersensitivity reactions to monoclonal antibodies (grade >= 3 National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v] 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
* Patients with a known history of severe interstitial lung disease or severe pneumonitis or active pneumonitis/pneumonia or pulmonary pathology that is not well controlled in the opinion of the treating physician and/or principal investigator (PI)
* Patients who have previously been treated with avelumab (or another PD1/PDL1 inhibitor) in combination with 5-azacytidine will be excluded
* Persisting toxicity related to prior therapy of grade > 1 NCI-CTCAE v 4.03; however, alopecia and sensory neuropathy grade =< 2 is acceptable
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent: a) subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible; b) subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses =< 10 mg or 10 mg equivalent prednisone per day; c) administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable
* Patients with organ allografts (such as renal transplant) are excluded
* Patients who are < 90 days post allogeneic stem cell transplant will be excluded; patients beyond 90 days post-allogeneic stem cell transplant with active uncontrolled graft versus host disease (GVHD) > grade 1 will be excluded; patients who are on a stable dose of immunosuppressive therapy (tacrolimus, cyclosporine, or other) for > 2 weeks will be eligible but those with recent increase in the immunosuppressive medication dose within last 2 weeks to control GVHD will not be included; Note: subjects may be using systemic corticosteroids or topical or inhaled corticosteroids post allogeneic stem cell transplant; patients requiring >= 1 mg/kg prednisone for GVHD management at the time of screening will not be eligible until the prednisone can be weaned to < 1 mg/kg; such patients should be monitored for at least 14 days and if no flare of GVHD requiring re-escalation of steroids or additional interventions for the GVHD they will be eligible
* Patients with symptomatic CNS leukemia or patients with poorly controlled CNS leukemia
* Active and uncontrolled disease/(active uncontrolled infection, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure New York Heart Association [NYHA] class III/IV, clinically significant and uncontrolled arrhythmia) as judged by the treating physician
* Patients with known human immunodeficiency virus seropositivity will be excluded
* Known to be positive for hepatitis B by surface antigen expression; known to have active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months)
* Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator
* All other significant diseases (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the investigator, might impair the subject's tolerance of trial treatment
* Patients unwilling or unable to comply with the protocol
* Pregnant or breastfeeding
* Known alcohol or drug abuse within the last 1 year
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines
* Acute promyelocytic leukemia (APL)
* Subject has a history of other malignancies prior to study entry, with the exception of: adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast; basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; previous malignancy confirmed and surgically resected (or treated with other modalities) with curative intent or completed definitive therapy (chemotherapy, radiation, others) for the malignancy at least 1 year prior to the date of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 2017 to February 2019
Groups:
- Treatment (Azacitidine, Avelumab): Patients receive azacitidine SC or IV over 10-40 minutes on days 1-7 or on days 1-5 and 8-9. Patients also receive avelumab IV over 60 minutes on days 1 and 14 for 4 courses (or until complete response) and on day 1 for subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Avelumab: Given IV
  Azacitidine: Given subcutaneous or IV
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Azacitidine, Avelumab)
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Azacitidine, Avelumab)
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 69 [22 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Complete Response (CR) + Partial Remission (PR) + Complete Remission with incomplete recovery (CRi) + Clinical Benefit. CR = normalization of peripheral blood (PB) and bone marrow (BM) with </= 5% BM blasts, PB granulocyte count >/= (1.0 x 10^9/L, and a platelet count >/= 100 x 10^9/L). PR = same as CR except presence of 6-15% marrow blasts, or 50% reduction if <15% at start of treatment. CRi meets all criteria for CR except for platelet recovery to >100 x 10^9/L and/or granulocyte count > (1.0 x 10^9/L). MLFS is BM with </= 5% BM blasts with no PB recovery. Hematologic Improvement is platelets increase by >/= 30 x 10^9/L untransfused (if <20 at pretherapy); or granulocytes increase by 100% and to >0.5 x 10^9/L (if lower than that pre-therapy); or hemoglobin increase by 2 g/dl; or transfusion independent; or splenomegaly reduction by > 50%; or monocytosis reduction by > 50% if pretreatment > 5 x 109/L, or BM or PB Blasts decrease by >/= 50%.
Time Frame: Up to 2 years
Population: Of the 19 participants registered, 17 participants were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Azacitidine, Avelumab)
Number analyzed (Participants) | 17
Participants | 4

2. Secondary Outcome: Disease-free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 1 year
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Azacitidine, Avelumab)
Number analyzed (Participants) | 17
Months | 8.2 [6.5 to 9.8]

3. Secondary Outcome: Overall Survival (OS)
Description: Distribution of OS will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Time Frame: Up to 1 year
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Azacitidine, Avelumab)
Number analyzed (Participants) | 17
Months | 4.7 [0.1 to 11.0]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Distribution of PFS will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Time Frame: Up to 1 year
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Azacitidine, Avelumab)
Number analyzed (Participants) | 17
Months | 3.2 [0.1 to 10.6]

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Treatment (Azacitidine, Avelumab)
All-Cause Mortality (participants affected / at risk) | 5/19
Serious Adverse Events (participants affected / at risk) | 18/19
Other Adverse Events (participants affected / at risk) | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Azacitidine, Avelumab) (N=19)
Anorectal Infection (Infections and infestations) | 2 (3)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 1 (1)
Death (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Neutropenic Fever (Infections and infestations) | 4 (4)
Fever (General disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infection (Infections and infestations) | 3 (6)
Lung Infection (Infections and infestations) | 6 (12)
Metabolism and Nutrition Disorder (Metabolism and nutrition disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 3 (4)
Skin Infection (Infections and infestations) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Azacitidine, Avelumab) (N=19)
Elevated Alanine Aminotransferase Increase (Investigations) | 2 (2)
Alkaline Phosphatase Increased (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 3 (3)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1)
Cardiac Troponin I Increase (Investigations) | 1 (1)
Cbills (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Fatigue (General disorders) | 4 (4)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Infusion Related Reaction (General disorders) | 4 (5)
Lymphocyte Count Decreased (Investigations) | 2 (2)
Mucosal Infection (Infections and infestations) | 1 (1)
Oral Mucositis (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (6)
Neutropenia (Investigations) | 2 (2)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1)
Platelet Count Decrease (Investigations) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (8)
White Blood Count Decreased (Investigations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT02953561/Prot_SAP_000.pdf